CLINICAL TRIAL: NCT06132282
Title: The Substance Use and Health Risk Intervention (SUHRI) for Justice-involved Youth
Acronym: SUHRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, DanicaKnight, Professor, Texas Christian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34DA048065 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: A technology-based application (administered via tablet) that addresses the interrelated topics of substance use and risky sex practices, within the context of personal relationships.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Substance Use and Health Risk Intervention (SUHRI) (Experimental): A technology-based application (administered via tablet) that addresses the interrelated topics of substance use and risky sex practices, within the context of personal relationships. This is the only arm for this clinical trial; and reflects pilot 2 only with accompanying IRB protocol.
  Interventions: Behavioral: Substance Use and Health Risk Intervention (SUHRI)

INTERVENTIONS:
Behavioral: Substance Use and Health Risk Intervention (SUHRI) — Technology-based intervention designed as 4 sessions administered on a tablet as a self-directed approach (requiring an onsite proctor) for addressing factors that increase risk for significant health problems. Topics such as SU and risky sex are important but often sensitive or difficult for juvenile justice staff to address in their role as probation officers.

SUMMARY:
This investigation will adapt and pilot test an integrated health risk-reduction and motivational enhancement intervention for Juvenile Justice (JJ) youth that will ultimately be (after full testing through a subsequent large-scale RCT) a sustainable intervention implemented within a JJ supervision/case management context to teach and facilitate positive, pro-social, and expected behaviors. The intervention will use graphical approaches to encourage introspection and problem identification, enhance self-regulation, improve analytical problem-solving skills, and promote healthy behaviors in two inter-related target areas: substance use and risky sex practices. Existing evidence-based intervention materials will be incorporated and delivered through a web-based application. Sessions will be self-directed (require minimal instruction/interaction assistance), and also include a service referral piece whereby youth are provided with a list of treatment and health agencies at the end of sessions that address specific topics. Research activities will be carried out in two pilot studies: (1) Intervention Adaptation and Feasibility and (2) Protocol Feasibility and Preliminary Efficacy Trial. In Pilot 1, intervention content will be adapted from existing evidence-based interventions so that it is developmentally appropriate for the target population and suitable for a web-based format (N = 30; 20 youth, 10 JJ staff). Pilot 2 will test a scaled-down version of an intervention efficacy trial, testing the web-based intervention using a 1-arm design whereby 60 enrolled youth (who meet eligibility requirements) from one juvenile probation department are enrolled to participate. This clinical trial submission, and the accompanying IRB protocol are based on pilot 2 only.

DETAILED DESCRIPTION:
A 1-arm design was used to examine preliminary efficacy of the adapted intervention. Youth aged 14 to 18 who are disposed to community supervision (deferred adjudication or probation) and meet eligibility requirements (1+ indicator of substance use, under community supervisions, English-speaking, no indication of suicide risk or thought disorder) were sampled from a large urban Texas juvenile probation department. Protocol administration was proctored by a TCU research assistant at a private space within a juvenile justice office or mutually agreed upon location of participant's choosing. Youth were asked to complete all assessments and participate in the 4 individualized technology-based intervention sessions where youth received information and engaged in decision making scenario-based games about substance use, sex risk practices, and related health-risk.

ELIGIBILITY:
Inclusion Criteria:

* on community supervision (e.g., deferred adjudication or probation), 1+ indicator of SU, English-speaking,

Exclusion Criteria:

* no indication of suicide risk or thought disorder

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Substance Use and Health Risk Intervention (SUHRI): A technology-based application (administered via tablet) that addresses the interrelated topics of substance use and risky sex practices, within the context of personal relationships.
  Substance Use and Health Risk Intervention (SUHRI): Technology-based intervention designed as 4 sessions administered on a tablet as a self-directed approach (requiring an onsite proctor) for addressing factors that increase risk for significant health problems. Topics such as SU and risky sex are important but often sensitive or difficult for juvenile justice staff to address in their role as probation officers.
  There is only one arm for this study, represented by pilot 2, and the accompanying IRB protocol
Period: Overall Study
Arm/Group | Substance Use and Health Risk Intervention (SUHRI)
Started | 40
Completed | 9
Not Completed | 31
Not completed — Lost to Follow-up | 31

BASELINE CHARACTERISTICS:
Groups:
- Substance Use and Health Risk Intervention (SUHRI): A technology-based application (administered via tablet) that addresses the interrelated topics of substance use and risky sex practices, within the context of personal relationships.
  Substance Use and Health Risk Intervention (SUHRI): Technology-based intervention designed as 4 sessions administered on a tablet as a self-directed approach (requiring an onsite proctor) for addressing factors that increase risk for significant health problems. Topics such as SU and risky sex are important but often sensitive or difficult for juvenile justice staff to address in their role as probation officers.
Arm/Group | Substance Use and Health Risk Intervention (SUHRI)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 15.76 [14 to 18]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  FEMALE | 8
  MALE | 27
  UNKNOWN | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 10
  More than one race | 3
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Service Initiation
Description: Number of Participants Who Initiated Substance Use or Health Services; obtained through client interviews.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use and Health Risk Intervention (SUHRI)
Number analyzed (Participants) | 40
Participants | 15

2. Primary Outcome: Service Initiation
Description: Number of Participants Who Initiated Substance Use or Health Services; obtained through client interviews.
Time Frame: Week 7
Population: those who completed the week 7 follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Substance Use and Health Risk Intervention (SUHRI)
Number analyzed (Participants) | 14
Participants | 4

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Substance Use and Health Risk Intervention (SUHRI)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Substance Use and Health Risk Intervention (SUHRI) (N=40)
hospitalization (General disorders) | 3
detention (Social circumstances) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT06132282/Prot_SAP_000.pdf